CLINICAL TRIAL: NCT01776645
Title: Compassion Training and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25883
Record Dates: First submitted 2013-01-15; First posted 2013-01-28 (Estimated); Results first posted 2013-12-16 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

ARMS (1):
- Compassion cultivation training (Experimental)
  Interventions: Behavioral: Compassion Cultivation Training Course

INTERVENTIONS:
Behavioral: Compassion Cultivation Training Course

SUMMARY:
The purpose of this study is to determine whether compassion training will improve the physical and psychological well-being of patients with chronic pain. The investigators also want to determine whether any benefit of compassion training in the patients "spreads" to significant others with whom the patient has a close relationship.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18+ and chronic pain for >6months
2. Pain over the last month
3. Ability to read, write, and converse in English
4. If being treated for pain condition, then stable treatment regimen.

For significant others:

1)18 years of age or older 2)Ability to read, write, and converse in English

Exclusion Criteria:

For patients and significant others:

1)Current or history of a psychological disorder that would interfere with study procedures, at the discretion of the researcher.

For patients only:

1. prior compassion meditation experience
2. on going legal action or disability claim
3. currently pregnant or planning to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Compassion Cultivation Training: Compassion Cultivation Training Course - Participants with Chronic Pain
- Significant Others Group: Significant others of the individuals with chronic pain undergoing the compassion cultivation training course
Period: Overall Study
Arm/Group | Compassion Cultivation Training | Significant Others Group
Started | 28 | 28
Completed | 14 | 14
Not Completed | 14 | 14

BASELINE CHARACTERISTICS:
Groups:
- Compassion Cultivation Training - Participants With Chronic Pa: Compassion Cultivation Training Course - Participants with Chronic Pain
- Significant Others Group: Significant Others of Participants with Chronic Pain
- Total: Total of all reporting groups
Arm/Group | Compassion Cultivation Training - Participants With Chronic Pa | Significant Others Group | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 24 | 50
  >=65 years | 2 | 4 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 49.61 (10.59) | 50.71 (12.59) | 50.16 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 7 | 31
  Male | 4 | 21 | 25
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change in Brief Pain Inventory
Description: Intensity - pain severity as measured by a 0 to 10 visual analogue scale. 0 = no pain, 10 = worst pain imaginable
Time Frame: Baseline and end of 9-week treatment protocol
Population: 2 participants excluded from analysis: 1 did not complete the final questionnaire battery, 1 reported no pain at baseline and thus could not be included as a patient with chronic pain
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Compassion Cultivation Training
Number analyzed (Participants) | 12
units on a scale | -1.46 (1.29)

2. Primary Outcome: Change in Chronic Pain Acceptance Questionnaire
Time Frame: Baseline and end of 9-week treatment protocol
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Change in Emotional Distress
Description: As assessed by the Hospital Anxiety and Depression Scale
Time Frame: Baseline and end of 9-week treatment protocol
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Overall Health and Well-being
Description: As assessed by Ryff's psychological well-being scales
Time Frame: Baseline and end of 9-week treatment protocol
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Compassion
Description: As assessed by Neff's Self-Compassion Scale
Time Frame: Baseline and end of 9-week treatment protocol
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Qualitative Measures
Description: Qualitative analysis of interviews
Time Frame: Baseline and end of 9-week treatment protocol
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Emotional Distress
Description: As Assessed by the PROMIS Anger Scale
Time Frame: Baseline and end of 9-week treatment protocol
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Emotional Distress
Description: As assessed by the PROMIS Social Isolation Scale
Time Frame: Baseline and end of 9-week treatment protocol
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Overall Health and Well-being
Description: As assessed by PROMIS Global Health Scale
Time Frame: Baseline and end of 9-week treatment protocol
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Compassion
Description: As assessed by Compassionate Love Scale adapted for close other
Time Frame: Baseline and end of 9-week treatment protocol
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Change in Compassion
Description: As assessed by Pommier's Compassion for Other's Scale
Time Frame: Baseline and end of 9-week treatment protocol
Reporting Status: Not Posted

12. Secondary Outcome: Change in Brief Pain Inventory
Description: Interference score - Interference as measured by a 0 to 10 numerical rating scale. 0 = does not interfere, 10 = completely interferes
Time Frame: Baseline to end of 9-week treatment protocol
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Compassion Cultivation Training
Number analyzed (Participants) | 12
units on a scale | -1.18 (1.94)

ADVERSE EVENTS:
Arm/Group | Compassion Cultivation Training | Significant Others Group
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 0/28 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes